CLINICAL TRIAL: NCT06628115
Title: Post-market Study of Cerament V/G in Foot Osteomyelitis
Brief Title: Post Market Study of Cerament V/G in Pedal Osteomyelitis
Acronym: Cerament 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: BONESUPPORT AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 339714
Record Dates: First submitted 2024-09-24; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Osteomyelitis - Foot
Keywords: osteomyelitis; antimicrobial; bone void filler; cerament
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Intervention Model Description: Case Series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cerament (Experimental): Cerament V/G implantation to forefoot or mid foot.
  Interventions: Device: cerament V or G

INTERVENTIONS:
Device: cerament V or G — Cerament V or G implantation into forefoot or mid foot bone, and 7-10 days of oral antibiotics.

SUMMARY:
The goal of this clinical trial is to look at the outcomes of patients who have had bone infection of their feet treated with a licensed antibiotic paste. The main question it aims to answer is:

• How does the bone infection heal in response to the antibiotic paste?

Participants will:

* Undergo standard surgery to remove dead bone and drain any pus.
* Antibiotic paste is injected directly into the middle of the bone at surgery. This is instead of receiving antibiotics directly into their bloodstream for 6 weeks.
* Recieve one week of tablet antibiotics.
* Visit clinic 1 month after surgery for a normal clinical appointment. After, a research team member will ask the participant a few questions. The participant will also have a foot x-ray, wound photograph and fill out a short questionnaire.
* Visit clinic 6 months and 12 months following the surgery. A research team member will ask the participant a few questions. The participant will also have a foot x-ray, wound photograph and fill out a short questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 18 years +
* Informed consent
* Operated on for foot sepsis with limb salvage intent.
* Positive bone biopsy from forefoot or midfoot or positive pus culture from exposed bone
* Adequate vascularity (1+ palpable pedal pulse, biphasic or triphasic ankle waveforms, or successful revascularisation procedure same admission)
* Compliant with offloading footwear and diabetic medication

Exclusion Criteria:

* Allergy or contraindication to gentamicin/vancomycin
* Life expectancy &amp <1 year
* Unable to make follow up appointments at study centre.
* Patients with necrotizing infections
* Gentamicin or vancomycin resistant organism
* Untreated peripheral arterial disease in angiosome of wound.
* Buerger's disease
* Vasculitides
* Systemic immunosuppressive therapy
* Pregnancy
* Breastfeeding
* Untreated thyrotoxicosis
* Mysathenia gravis
* Calcium metabolism disorder
* Patients taking metformin with estimated glomerular filtration rate (eGFR) > 30ml/min/1.72m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from clinical or radiological osteomyelitis in the same or adjacent bone (recorded as yes or no) | 12 months post-implantion
  Clinical osteomyelitis:
  positive bone biopsy in the setting of bone necrosis or purulent fluid containing pathogenic organisms emanating from exposed bone end.
  Radiological osteomyelitis:
  osteolysis or periosteal reaction on radiograph in affected or adjacent bone(s).
  This is checked at each follow up visit, at 1, 6 and 12 months post-implantation.

SECONDARY OUTCOMES:
Surgical site infection requiring further course of antibiotics (recorded as yes or no) | 12 months post-implantion
  If there is infection at the surgical site, requiring a further course of antibiotics, this will be recorded.
Major or minor amputation of study limb (recorded as yes or no with amputation details) | 12 months post-implantion
  If major or minor amputation of study limb occurs, this will be recorded.
Serious adverse events related to Cerament V/G (number and type of event are recorded) | 12 months post implantation
  A serious adverse event (SAE) refers to any expected or unexpected adverse event, related to ceramist, that results in any of the following outcomes: death, a life-threatening adverse event, requires inpatient hospitalisation (not required as part of the treatment) or prolongation of existing hospitalisation, a persistent or significant disability or incapacity, or cancer, or a congenital anomaly or birth defect.
Total treatment costs for osteomyelitis (total cost is calculated in GB pounds) | 12 months post-implantation
  Treatment costs will be collected through the use of a Client Service Research Inventory focussed on surgical, community and further treatment costs over a 12 month follow up. These will be recorded by the patient as they occur and checked at each visit and cross reference with hospital medical records.
Wound healing (recorded as yes or no) | 12 months post-implantation
  Wound is considered healed at 100% epithelialisation. This is checked at each follow up visit, at 1, 6 and 12 months post-implantation.
Wound area (measured in cm^2) | 12 months post-implantation
  Wound area is measured at each follow up visit, at 1,6 and 12 months post-implantation, using an app called Imito measure.
Quality of life (measured using the EQ-5D questionnaire) | 12 months post-implantation
  Quality of life is measured using the EQ-5D questionnaire. It is conducted at each follow up visit, at 1, 6 and 12 months post-implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Ankur Thapar, Principal Investigator — Mid and South Essex NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Yes
Anonymised outcome data for primary and secondary endpoints to 12 months will be made available for IPD meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 01/11/2026 to 1/11/2036
Access Criteria: Ankur Thapar
URL: http://www.aru.ac.uk/people/ankur-thapar

REFERENCES:
- [Background] Venkateswaran V, Tiruveedhula M, Edwards J, Dindyal S, Mulcahy M, Thapar A. Antibiotic Eluting Bone Void Filler Versus Systemic Antibiotics For Pedal Osteomyelitis. J Foot Ankle Surg. 2025 Jan-Feb;64(1):30-35. doi: 10.1053/j.jfas.2024.08.010. Epub 2024 Aug 23. PMID 39182821